CLINICAL TRIAL: NCT00322075
Title: Comparison of Glycaemic Fluctuations During 3 Days Subcutaneous Continuous Monitoring in Patients With Basal Substitution Human Insulin NPH vs Insuline Glargine
Brief Title: LANCGMS - Lantus Continuous Glucose Monitoring Subcutaneous
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_00722; EudraCT # : 2006-000122-31
Record Dates: First submitted 2006-04-27; First posted 2006-05-04 (Estimated); Last update posted 2007-09-12 (Estimated); Status verified 2007-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

INTERVENTIONS:
Drug: insulin glargine

SUMMARY:
Comparison of incidence of hypoglycaemic events and glycaemic fluctuations in diabetic patients with basal substitution with NPH insuline versus insuline glargine. Evaluation of HbA1c, FBG (Fasting Blood Glucose), BMI (Body Mass Index), dose of insulin, ratio of basal and prandial insulin, satisfaction with treatment, incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetes Mellitus Type 1 and Diabetes Mellitus Type 2 with HbA1c 6% and more with more than 2 confirmed hypoglycaemic events (glycaemia less than 3,3 mmol/l) during last year

Exclusion Criteria:

* Diabetic ketoacidosis
* Any other severe disease
* Pregnancy or fertile female without contraception
* Alcohol/drug abuse, selected prohibited concomitant medication
* Nightshift work

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2006-04; Study Completion 2006-11

PRIMARY OUTCOMES:
3 days continual glycaemic profile fluctuation
occurrence of adverse events
HbA1c
FBG
BMI
total daily dose of insulin and ratio of doses of basal/prandial insulines
patients´satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Priborska, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Prague, Czechia